CLINICAL TRIAL: NCT02188420
Title: Effect of Different Interpulse Intervals of Paired Associative Stimulation on Cortical Excitability in People With Chronic Stroke
Brief Title: Finding an Optimal Latency for Paired Associative Stimulation in People With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 1406M51743
Record Dates: First submitted 2014-06-30; First posted 2014-07-11 (Estimated); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Stroke
Keywords: PAS; TMS; Stroke; Paired Associative Stimulation; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- N20-3ms, N20-5ms, N20+100ms, N20-7ms (Experimental): Transcranial Magnetic Stimulation will be applied to the primary motor cortex at the interstimulus interval of ("Latency" - 3ms) where "latency" refers to the amount of time for the arrival of a sensory evoked potential as determined by EEG. Wash out period of 1 week then next level will be applied
  Interventions: Device: Transcranial Magnetic Stimulation will be applied to the primary motor cortex at the interstimulus interval of ("Latency" - 3ms)
- N20-5ms, N20-3ms, N20-7ms, N20+100ms (Experimental): Transcranial Magnetic Stimulation will be applied to the primary motor cortex at the interstimulus interval of ("Latency" - 5ms) where "latency" refers to the amount of time for the arrival of a sensory evoked potential as determined by EEG. Wash out period of 1 week then next level will be applied
  Latency minus 7ms Wash out period of 1 week Latency plus 100ms Active comparator
  Interventions: Device: Transcranial Magnetic Stimulation will be applied to the primary motor cortex at the interstimulus interval of ("Latency" - 5ms)
- N20-7ms, N20-5ms, N20-3ms,N20+100ms (Experimental): Transcranial Magnetic Stimulation will be applied to the primary motor cortex at the interstimulus interval of ("Latency" - 7ms) where "latency" refers to the amount of time for the arrival of a sensory evoked potential as determined by EEG. Wash out period of 1 week then next level will be applied
  Interventions: Device: ranscranial Magnetic Stimulation will be applied to the primary motor cortex at the interstimulus interval of ("Latency" - 7ms)
- N20-3ms, N20+100ms, N20-5ms, N20-7ms (Active Comparator): Transcranial Magnetic Stimulation will be applied to the primary motor cortex at the interstimulus interval of ("Latency" - 100ms) where "latency" refers to the amount of time for the arrival of a sensory evoked potential as determined by EEG. Wash out period of 1 week
  Interventions: Device: Transcranial Magnetic Stimulation Time 100ms

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation will be applied to the primary motor cortex at the interstimulus interval of ("Latency" - 3ms) — Transcranial Magnetic Stimulation will be applied to the primary motor cortex at the interstimulus interval of ("Latency" - 3ms) where "latency" refers to the amount of time for the arrival of a sensory evoked potential as determined by EEG.
  Other Names: TMS; Magstim
  Arms: N20-3ms, N20-5ms, N20+100ms, N20-7ms
Device: Transcranial Magnetic Stimulation will be applied to the primary motor cortex at the interstimulus interval of ("Latency" - 5ms) — Transcranial Magnetic Stimulation 5ms
  Other Names: TMS
  Arms: N20-5ms, N20-3ms, N20-7ms, N20+100ms
Device: ranscranial Magnetic Stimulation will be applied to the primary motor cortex at the interstimulus interval of ("Latency" - 7ms) — Transcranial Magnetic Stimulation 7ms
  Other Names: TMS
  Arms: N20-7ms, N20-5ms, N20-3ms,N20+100ms
Device: Transcranial Magnetic Stimulation Time 100ms — Active Compator
  Other Names: TMS
  Arms: N20-3ms, N20+100ms, N20-5ms, N20-7ms

SUMMARY:
After a stroke, there is an exaggerated inhibitory influence from the non-stroke hemisphere to the stroke hemisphere. Brain stimulation using repetitive transcranial magnetic stimulation (rTMS) to the non-stroke hemisphere can decrease this inhibition. Paired Associative Stimulation (PAS) may be a more effective way to produce this same inhibition, as shown in healthy subjects. However, it is not known whether this will translate to people with stroke. PAS consists of a peripheral nerve stimulus paired a short time later with a cortical stimulus to change the excitability within the brain. Thus the investigators will apply PAS to people with stroke, but the investigators need to first determine the most effective interpulse interval (IPI) between the peripheral and cortical stimuli. Our research question is which of three different IPIs is most effective in changing the excitability of the brain.

The purpose of this study is to determine the optimal IPI between a peripheral nerve pulse and a cortical stimulus that will be most effective in changing excitability of the brain in people with chronic stroke. The investigators hypothesize that the cortical excitability of the nonstroke hemisphere will be most inhibited with the latency-5ms condition.

DETAILED DESCRIPTION:
Numerous PAS studies have been done in healthy subjects and all have been done safely. The proper interpulse interval in healthy individuals between the peripheral nerve stimulus and the cortical stimulus is known to be "latency-5ms." However, this may be different in individuals with stroke.

Specific Aim: what is the optimal interpulse interval to achieve the maximum inhibitory effect in the nonstroke hemisphere?

We will recruit three subjects with chronic stroke. Electroencephalography (EEG) will be used to determine the latency between the peripheral nerve stimulus and the sensory evoked potential in each subject. We will then assess the following IPIs on each subject in a random order: "latency" - 3ms, -5ms and -7ms. There will be a fourth condition of "latency" + 100ms (known to have no effect) to be used as a control. The washout period will be at least one week between each of these conditions.

The optimal IPI will be determined from these tests by comparing single pulse transcranial magnetic stimulation (TMS) measures for cortical excitability. Prior to each treatment, each subject will receive 20 single pulse cortical stimuli to serve as pretest data. The post tests for each condition will consist of 20 single pulse cortical stimuli at 0, 5, 10, 15, 30, 45 and 60 minutes after the PAS condition. Data analysis will consist of a single-subject analysis with the two standard deviation bandwidth method of each post-test compared to pre-test.

We hypothesize that there will be no adverse advents and that this optimal IPI will be "latency"-5ms.

ELIGIBILITY:
Inclusion Criteria:

* stroke (ischemic or hemorrhagic) of greater than 6 months duration
* impairment in the paretic hand
* over 18 years old
* male or female
* on mini mental status exam must have score of 22 or higher
* must have elicitable motor evoked potential (MEP)

Exclusion Criteria:

* seizure within the past two years
* receptive aphasia
* epileptogenic medication
* major psychiatric disorder
* other interfering comorbidities
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate Frost, MS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Clinical and Translational Science Institute, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were no significant events or excluded participants prior to being assigned an intervention order
Groups:
- Group 1: Randomized Sequence 1) N20-3ms, N20-5ms, N20+100ms, N20-7ms
- Group 2: Randomized Sequence 2) N20-3ms, N20+100ms, N20-5ms, N20-7ms
- Group 3: Randomized Sequence 3) N20-7ms, N20-5ms, N20-3ms, N20+100ms
- Group 4: Randomized Sequence 4) N20-5ms, N20-3ms, N20-7ms, N20+100ms
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: This is a cross-over study; all participants completed all four treatment arms.
Arm/Group | All Study Participants
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Cortical Excitability Using Single TMS Pulses
Description: Assess average size of 20 motor evoked potentials via electromyography (EMG) signal resulting from single TMS pulses to the motor cortex. Measurements taken before and after paired associative stimulation treatment at each session.
Time Frame: Change from pretest (immediately prior to PAS application) to posttest which will occur over the 60 minutes that follow PAS application.
Measure: Mean (Standard Deviation); unit: Log10(microvolts)
Groups:
- Latency Minus 3ms: Transcranial Magnetic Stimulation will be applied to the primary motor cortex at the interstimulus interval of ("Latency" - 3ms) where "latency" refers to the amount of time for the arrival of a sensory evoked potential as determined by EEG.
  Transcranial Magnetic Stimulation (Magstim)
- Latency Minus 5ms: Transcranial Magnetic Stimulation will be applied to the primary motor cortex at the interstimulus interval of ("Latency" - 5ms) where "latency" refers to the amount of time for the arrival of a sensory evoked potential as determined by EEG.
  Transcranial Magnetic Stimulation (Magstim)
- Latency Minus 7ms: Transcranial Magnetic Stimulation will be applied to the primary motor cortex at the interstimulus interval of ("Latency" - 7ms) where "latency" refers to the amount of time for the arrival of a sensory evoked potential as determined by EEG.
  Transcranial Magnetic Stimulation (Magstim)
- Latency Plus 100ms: Transcranial Magnetic Stimulation will be applied to the primary motor cortex at the interstimulus interval of ("Latency" + 100ms), known to have no effect, where "latency" refers to the amount of time for the arrival of a sensory evoked potential as determined by EEG.
  Transcranial Magnetic Stimulation (Magstim)
Arm/Group | Latency Minus 3ms | Latency Minus 5ms | Latency Minus 7ms | Latency Plus 100ms
Number analyzed (Participants) | 3 | 3 | 3 | 3
Log10(microvolts) | -.07667 (0.06184) | 0.11 (0.06164) | -.05667 (0.2625) | .1233 (0.15173)

ADVERSE EVENTS:
Arm/Group | Latency Minus 3ms | Latency Minus 5ms | Latency Minus 7ms | Latency Plus 100ms
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes